CLINICAL TRIAL: NCT03448289
Title: Use of a Reproductive Life Planning Tool at the Pediatric Well-Baby Visit With Postpartum Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Rachel N Caskey, Chief, Division of Academic Internal Medicine, University of Illinois at Chicago
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2017-1009; 1R03HS025265-01A1 (AHRQ)
Record Dates: First submitted 2018-02-07; First posted 2018-02-28 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Postpartum Period; Contraception Behavior; Women's Health; Primary Health Care
Keywords: Postpartum; Contraception
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Intervention Model Description: The control group will be enrolled during phase 1 (first 4 months) prior to the introduction of the intervention. After enrollment of the control group, a 6-week washout period prior to phase 2 (intervention) will ensure women are not enrolled into both arms of the study.
Who Masked: Participant
Masking Description: Because we are studying health behaviors, we cannot share the specific aims of the study with control group participants as this could bias behavior. The control group participants will be told that this is a study monitoring women's general health care experiences at UIH.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): This group will not receive the RLPT.
- Intervention (Experimental): This group will receive the RLPT.
  Interventions: Behavioral: RLPT

INTERVENTIONS:
Behavioral: RLPT — The Reproductive Life Plan Tool (RLPT) will be self-administered. Pediatricians will use the RLPT to assess women's need for well-woman primary care.
  Arms: Intervention

SUMMARY:
Improved access to timely health care and contraception in the postpartum (PP) period is needed to reduce unintended pregnancies and help women achieve desired birth spacing. While the routine 6-week visit has historically been considered the place for women to discuss and receive contraception, many women, particularly low-income women, do not attend the postpartum visit. A novel approach to increasing receipt of PP care and contraception is the adoption of a reproductive life planning tool. Explorations of the use of a self-administered Reproductive Life Plan Tool (RLPT) by pediatricians in the context of the Well-Baby Visit (WBV) with postpartum mothers, holds great promise.

The objective of this study is to determine whether use of a simple self-administered Reproductive Life Plan Tool at the 2-month WBV increases the proportion of postpartum women receiving woman's health care and contraception at 6-months PP, compared to women not exposed to such an intervention. The two specific aims of the project are: 1) To determine if introducing a self-administered Reproductive Life Planning Tool (RLPT) with postpartum mothers during the 2-month WBV will increase the proportion of women receiving a well-woman primary care health visit by 6 months postpartum; and if introducing a self-administered Reproductive Life Planning Tool (RLPT) will increase utilization rates of contraception by 6 months postpartum. 2) To assess patient-, provider-, and systems-level barriers and facilitators to integrating a self-administered Reproductive Life Planning Tool (RLPT) designed to facilitate referral of postpartum women for primary well-woman care in the context of a pediatric clinic.

The investigators hypothesize that exposure to a self-administered RLPT combined with a conversation with a pediatrician during a 2-month WBV will increase use of well-woman primary health care during the postpartum period as well as receipt of contraception, by 6-months postpartum. If successful, the results of this study have great potential to inform clinical and public health practice to increase women's use of health care and contraception in the postpartum period.

DETAILED DESCRIPTION:
Specific Aims Aim I. To determine if introducing a self-administered Reproductive Life Planning Tool (RLPT) with postpartum mothers during the 2-month WBV will increase the proportion of women receiving a well-woman primary care health visit by 6 months postpartum.

Aim Ia. To determine if introducing a self-administered Reproductive Life Planning Tool (RLPT) with postpartum mothers during the 2-month WBV will increase utilization rates of contraception by 6 months postpartum.

Aim II: To assess the extent of system adoption as well as patient-, provider-, and systems-level barriers and facilitators to integrating a self-administered Reproductive Life Planning Tool designed to facilitate referral of postpartum women for primary well-woman care within the context of a pediatric clinic.

Study Design and Intervention This is a single-site system-level pilot study to measure the impact of a self-administered RLPT during the 2-month WBV on PP women's subsequent receipt of primary health care and contraception, compared to usual care. To facilitate women's uptake of a referral for well-woman primary care, mothers will be offered the opportunity to schedule a well-woman visit on the same day as their infant's next WBV or the first available visit if the participant needs more immediate care. This study will have two phases: phase 1 is enrollment of a control or baseline group, followed by a washout period; phase 2 is enrollment of the intervention group (intervention).

During phase 2 (intervention), the self-administered RLPT will be implemented in the Child and Youth Center (CYC, the general pediatric clinic) and the Primary Care Adolescent and Child Clinic (PCAC) at UIH with all PP women bringing infants for the 2-month WBV. The intervention leverages an existing system designed to screen all PP women (through 6-months) for depression.

During the WBV, physicians will review the information provided by the woman on the RLPT about general health, reproductive plans, and use of contraception. The pediatrician will use the RLPT to initiate a brief conversation with mothers about the need for a referral for well-woman primary care. The investigators will create a referral process to the UIH Primary Care Plus clinic (internal medicine) through the electronic medical record. At the close of the WBV, if the mother desires a referral the pediatrician can request the referral during the infant's check-out process. Research staff will routinely review all referral needs and initiate scheduling based on the mother's preference. Mothers will be asked for a preference of the next available appointment or an appointment on the same day as the infant's next WBV. For women who desire their health care visit on the same day as their infant's next WBV (the 4-month visit), a research assistant will schedule both visits on the same day. To the extent possible, the mother's appointment will be earlier the same day (ideally 2 hours before) of the infant's scheduled visit, to promote attendance.

Participant Recruitment into the Research Study: The intervention is planned as a system-level intervention, thus, all women whose infants are scheduled for a 2-month WBV during the intervention period will have the opportunity to be exposed to the RLPT intervention. On study recruitment days (randomly selected half-days during phase 2), women whose infants are scheduled for a 2-month WBV will be approached by a research assistant (RA) who will screen for eligibility. Recruitment into the study will occur before, during or after the WBV, baseline surveys will be completed during or after the WBV to avoid biasing women's responses on the RLPT, which is administered prior to the WBV. If a woman is eligible and interested in participating, the subject will be consented and asked to complete a baseline survey.

After consent is obtained, the RA will cross-check the participant list using a secure network on a tablet device to ensure that the woman is not already enrolled. Each RLPT will be linked to the infant by medical record number and date of birth. Limited physician characteristics (male/female, trainee/faculty) will be recorded; no physician names will be collected. The RLPTs for women who are consented and enrolled in the study will remain intact and all data will be collected from the tool and linked to the enrolled mother. The RLPTs for women who are not enrolled into the study will be de-identified after the Edinburgh tool is scanned by removing and shredding the patient sticker so no identifying information remains on the form. This will allow the investigators to calculate clinic-specific adoption rates and examine the extent to which provider and system characteristics, such as the type of physician (e.g., attending versus resident), demographic characteristics of the physician (e.g., sex), and clinic operational factors (e.g., morning versus afternoon clinic; day of the week), influences adoption of the intervention.

Consent for Intervention Group: Informed consent will be obtained for: 1) a baseline survey; 2) a phone survey at 6 months PP; and 3) access to a woman's medical records to document receipt of health care services. Women will be will reimbursed for their time with gift cards [$10 at baseline and $10 at follow-up (6-month WBV)]. The RA will log the recruitment process, including number of women approached and if women accepted or refused, participation.

Selection of Control Group: The control group will be enrolled during phase 1 (first 4 months) using similar procedures as the Intervention Group, but prior to the introduction of the intervention. After enrollment of the control group, a 6-week washout period prior to phase 2 (intervention) will ensure women are not enrolled into both arms of the study.

Pediatrician Training: Pediatricians (faculty and resident physicians) will all receive a 1-hour formal training on using the RLPT prior to the start of the study, offered at three different times to accommodate physician schedules. Research staff will touch-base with pediatricians weekly during the first 4 weeks of the study, and monthly thereafter, to answer questions and encourage consistent provider use of the tool. The researchers will schedule a 'refresher' training 3 months after the start of the study to reinforce appropriate use of the tool. During the training, physicians will be instructed on how to start a conversation with women, what to document on the tool, and how to initiate a referral if needed. Physicians are not expected to provide contraceptive counseling to mothers, only to engage women in a discussion about their health care needs. An information sheet about the study will be given to all pediatric providers who are trained.

Sample: This pilot study will enroll at least 50 women per group. This sample size will provide a stable estimate of the intervention's effect on primary care receipt by 6 months postpartum for power calculations for a larger, subsequent study of intervention effectiveness.

Data Sources and Collection Surveys of Women: All participants will complete a baseline survey (English or Spanish) at the time of enrollment in the study (during or after the WBV) and will receive a phone call at 6 months PP for the follow-up survey. During the baseline survey, in addition to demographic information, women will be asked about their general health status and health behaviors, and current contraception type and use. Those in intervention arm will be asked about their experience completing the RLPT during the WBV, referral to well-woman primary care (if applicable). For the follow-up survey the researchers will try to reach each participant as close to 6 months as possible, but no later than 9 months PP. Structured phone interviews with women will include questions from the following domains: 1) use of health care services; 2) use and type(s) of contraception; and 3) known pregnancy status. The intervention group interviews will also include experience completing the RLPT during the WBV; and, the process of getting care (for those who chose to do so) (SA II). To verify RLPT exposure at the individual level, the RLPT tool will be linked to the mother using the patient sticker placed on the tool.

Medical Records: Medical records will be reviewed at baseline and at 6 months PP to determine receipt of health care services and contraception. The investigators recognize that some women may receive additional health care outside the UIC system; for this group, the researchers will not be able to confirm medical visits outside the UIC system.

Focus Groups with Providers: The investigators will conduct two in-depth qualitative focus groups with physicians (residents and faculty) after the intervention is complete during study year 2. The focus group guide will include questions from the following domains: 1) Experience implementing the RLPT; and, 2) barriers and facilitators to implementation of RLPT (SA II). In addition, study investigators will keep a running log of barriers and facilitators experienced throughout the intervention implementation period.

Data Management All survey data will be directly entered into REDcap web-based data capture screens that will be programmed and tested prior to the study. Data will be imported to SAS for analysis. Variables will be merged across time point by study ID and cleaned and recoded. Focus groups will be recorded, transcribed, and uploaded to DeDoose qualitative analysis software. Completion of the Grey Box (physician section of the tool) will be a measure of provider "adoption" of the intervention; completion rates will be tracked by comparing completed forms with completed clinic visits for 2-month WBVs. Completed clinic visit data are available in the existing medical record scheduling system.

Analysis Specific Aim I and Ia: Baseline characteristics will be assessed for equivalency across groups using chi-square tests for categorical and t-tests for continuous variables. Unbalanced characteristics will be adjusted for in further analyses. An intent-to-treat analysis will be performed for SA I and Ia. A crude relative risk (RR) and risk difference (RD) will be calculated with 95% confidence intervals to estimate the effect of the intervention on primary outcomes. If adjustment is needed for covariates, RRs and RDs will be estimated using the average marginal predictions from a fitted logistic regression model with the following form:41

logit(y) = β0 + β1x1 + β2x2 + …+ βkxk , where: y = SA 1: Woman's primary care visit by 6 months (1 = Yes/0 = No) SA 1a: Use of contraception at 6 months (1 = Yes/0 = No) x1 = RLPT Intervention (1 = Intervention/0 = Control) x2 - xk = Unbalanced covariates

Although the findings of this study will reflect the experiences of low-income women at one large medical center in Chicago, the experiences are likely to be relevant to those of many low-income women. While a hospital outpatient clinic is a unique health care setting, the experience of having a pediatrician discuss new mothers' health needs and refer mothers for their own care is likely to be similar across pediatric practices. This study will add to the emerging literature related to a dual care focus for mother and infant. If this intervention is successful, this work will provide evidence of the feasibility of introducing a system-level intervention related to women's health into pediatric practice. This information can inform changes in payment and policy to support the ability of pediatricians to discuss women's health needs and facilitate referral with mothers at their infants' WBV, with the ultimate goal of increasing women's use of primary care and PP contraception, preventing rapid repeat and unintended pregnancies, and ultimately decreasing adverse pregnancy outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum women 15-49 years
* Present with infant for a 2-month WBV at the UIC CYC or PCAC
* Receive healthcare at UIC
* Speak English or Spanish

Exclusion Criteria:

* Pregnant
* < 15 years or > 49 years of age
* Receive healthcare outside the UIC system
* Do not speak English or Spanish

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Postpartum women
Enrollment: 129 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2019-09-29 (Actual); Study Completion 2019-09-29 (Actual)

PRIMARY OUTCOMES:
Change in receipt of primary care services - self report | 2-months and 6-months Postpartum (baseline and 4-months from baseline data collection)
  Change in receipt of primary care services will be ascertained by self-report on the 2-month and 6-month Postpartum interview.
Change in receipt of primary care services - EMR review | 2-months and 6-months Postpartum (baseline and 4-months from baseline data collection)
  Change in receipt of primary care services will be ascertained by electronic medical record review at 2-months and 6-months Postpartum. Evidence of a visit from either source (self-report or EMR review) will be counted as receipt.

SECONDARY OUTCOMES:
Contraception utilization | 2-months and 6-months Postpartum (baseline and 4-months from baseline data collection)
  Change in contraception utilization will be assessed using the 2-month baseline survey and the 6-months Postpartum interview.
Participant feasibility and acceptability | The last half of Year 2
  Patient barriers and satisfaction data will be gathered from the RLPT and surveys. System adoption will be defined as the number of completed RLPT forms clinic-wide during the intervention (for enrollees and non-enrollees) divided by the total number of eligible visits during that time period, which will be ascertained through the clinic's scheduling database. Women's perceptions of feasibility and acceptability will be derived through the survey data and will be analyzed by other key covariates.
Provider feasibility and acceptability | The last half of Year 2
  System adoption statistics will be shared with providers prior to focus groups, allowing them to elaborate on these findings. Qualitative focus group data from providers will be coded according to domains and analyzed for emergent themes related to feasibility and acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Caskey, MD, MAPP, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Caskey RN, Olender SE, Zocchi A, Bergo CJ, Uesugi KH, Haider S, Handler AS. Addressing Women's Health Care Needs During Pediatric Care. Womens Health Rep (New Rochelle). 2021 Jul 9;2(1):227-234. doi: 10.1089/whr.2021.0016. eCollection 2021. PMID 34318292
- [Derived] Yonemoto N, Nagai S, Mori R. Schedules for home visits in the early postpartum period. Cochrane Database Syst Rev. 2021 Jul 21;7(7):CD009326. doi: 10.1002/14651858.CD009326.pub4. PMID 34286512

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-25): https://cdn.clinicaltrials.gov/large-docs/89/NCT03448289/Prot_SAP_000.pdf